CLINICAL TRIAL: NCT01015820
Title: Detectable Early Increase in Blood Flow (EIBS) in the Duodenum in Patients With Pancreatic Cancer
Brief Title: Early Increase in Blood Flow (EIBS) in the Duodenum in Patients With Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Northwestern University (Other); National Cancer Institute (NCI) (NIH); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Principal Investigator, Michael Wallace, M.D., Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 09-002596; R01CA128641 (NIH); R01CA156186 (NIH); R01EB003682 (NIH); U01CA111257 (NIH); CBET-1240416 (Other Grant/Funding Number: National Science Foundation)
Record Dates: First submitted 2009-11-12; First posted 2009-11-18 (Estimated); Results first posted 2014-07-02 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Duodenum; Spectroscopy; Fiberoptic probe; 4D-ELF
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cancer group (Experimental): Participants in this group had pathologically confirmed pancreatic adenocarcinoma. They received an EGD with EUS. During the EUS, blood flow was measured in the duodenum with the 4D-ELF device.
  Interventions: Procedure: EGD with EUS; Device: 4D-ELF
- Control group (Other): Participants in this group were without pancreatic adenocarcinoma. Participants in the control group received an EGD with EUS for the indication of abdominal pain. During the EUS, blood flow was measured in the duodenum with the 4D-ELF device.
  Interventions: Procedure: EGD with EUS; Device: 4D-ELF

INTERVENTIONS:
Procedure: EGD with EUS — EUS was performed in order to measure blood flow in duodenum.
Device: 4D-ELF — During the EUS, blood flow was measured in the duodenum with the 4D-ELF device.

SUMMARY:
Pancreatic cancer is the fourth leading cause of cancer death in the United States and is associated with a poor prognosis. The average life expectancy after diagnosis is approximately 5 to 8 months. At present, successful surgical resection is the only curative therapy that can improve long-term survival. However, it can be achieved only when a tumor is detected at an early stage. Unfortunately, due to non-specific symptoms associated with pancreatic cancer, it is commonly detected in the later stages of the disease.

The investigators hypothesized that pancreatic cancer could be detected by measuring the changes in the early increase in blood supply (EIBS) found in the surrounding normal-appearing duodenal tissue. The investigators tested a device called Four-dimensional Elastic Light-Scattering Fingerprinting (4D-ELF). The device used in this study is considered investigational, which means it has either not been approved by the Food and Drug Administration (FDA) for routine clinical use or for the use described in this study. However the FDA allowed the use of this device in this research study.

DETAILED DESCRIPTION:
According to field effect theory, by detecting microvasculature changes in the early increase of blood supply in the surrounding tissue neoplastic lesions can be identified from a distance.

The objective of this study was to determine the feasibility and efficacy of a fiberoptic probe containing novel Polarization Gating Spectroscopy (PGS) technology to identify patients with pancreatic adenocarcinoma (PAC) by field effect theory. EIBS markers, deoxyhemoglobin concentration (DHb), and average blood vessel radius (BVR) were evaluated in patients with PAC versus controls.

During the subjects' esophagogastroduodenoscopy (EGD) with upper endoscopic ultrasound (EUS), the new optic probe was inserted inside the endoscope and advanced to the tip of the endoscope prior to the scope being withdrawn. As the scope was withdrawn, the light optic probe was used to examine approximately 5 sections of the small bowel: 1) directly on the ampulla, 2) approximately 5 mm proximal from the ampulla, 3) approximately 5 mm distal from the ampulla, 4) 1 cm proximal from the ampulla, and 5) 1 cm distal from the ampulla. Spectroscopy measurements were obtained four times in each of these five peri-ampullary locations. The rest of the EGD and upper EUS endoscopy procedures were then completed as clinically indicated. During the procedure, all visualized mucosal abnormalities were recorded and photographed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Informed written consent.
* Patient scheduled for previously planned EGD with upper EUS
* Patients with known adenocarcinoma of the pancreas included in the cancer group
* Patients with abdominal imaging studies (e.g., CT abdomen or MRI abdomen) negative for malignancy in past 5 years included in the control group.

Exclusion Criteria:

* Unable to obtain biopsy specimen or fine-needle aspiration results of the pancreas lesion (e.g., coagulation disorder, inadequate sample)
* Presence of malignant lesion in the pancreas or duodenum other than pancreas adenocarcinoma (e.g., neuroendocrine tumor, gastrointestinal stromal tumor)
* Known familial disorder with high risk of pancreas cancer development (e.g., familial adenomatous polyposis syndrome, hereditary non-polyposis colorectal cancer syndrome, juvenile polyposis syndrome)
* Significant family history of pancreatic cancer (at least one first degree relative with pancreatic cancer)
* Presence of premalignant lesions (e.g., duodenal adenoma, pancreas intraductal papillary mucinous neoplasm)
* Active visible inflammation/ulcer in the stomach or the duodenum
* Patients with known chronic pancreatitis were excluded from cancer group. Chronic pancreatitis patients were allowed to be included in the control group only.
* Known pregnancy or sexually active females of childbearing age who are not practicing an accepted form of birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael B. Wallace, MD MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

REFERENCES:
- [Result] Patel M, Gomes A, Ruderman S, Hardee D, Crespo S, Raimondo M, Woodward T, Backman V, Roy H, Wallace M. Polarization gating spectroscopy of normal-appearing duodenal mucosa to detect pancreatic cancer. Gastrointest Endosc. 2014 Nov;80(5):786-93.e1-2. doi: 10.1016/j.gie.2014.03.031. Epub 2014 May 24. PMID 24861243

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 37 patients were enrolled in the study. Of these, 5 patients with neuroendocrine tumors and 2 patients with duodenal anatomy limiting the use of the probe were excluded because of screen failure.
Groups:
- Cancer Group: Participants in this group had pathologically confirmed pancreatic adenocarcinoma. They received an esophagogastroduodenoscopy (EGD) with endoscopic ultrasound (EUS). During the EUS, blood flow was measured in the duodenum with the Four-dimensional Elastic Light-Scattering Fingerprinting (4D-ELF) device.
Period: Overall Study
Arm/Group | Cancer Group | Control Group
Started | 15 | 15
Completed | 14 | 15
Not Completed | 1 | 0
Not completed — Suboptimal measurements | 1 | 0

BASELINE CHARACTERISTICS:
Population: Among the 15 participants in the cancer group, 1 participant was excluded from the final analysis due to suboptimal measurements. Therefore 14 participants in the cancer group and 15 participants in the control group were included in the baseline analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cancer Group | Control Group | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (10) | 63 (11) | 67 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 11 | 9 | 20
Region of Enrollment [Number; unit: participants]
  United States | 14 | 15 | 29

OUTCOME MEASURES:

1. Primary Outcome: Deoxyhemoglobin Concentration (DHb)
Description: Deoxygenated hemoglobin is the form of hemoglobin without the bound oxygen. It serves as a marker for early increase of blood supply (EIBS). DHb concentration was determined spectroscopically from five peri-ampullary locations.
Time Frame: Completion of study procedure (endoscopic ultrasound), approximately 30 minutes from procedure initiation
Population: Among the 15 participants in the cancer group, 1 participant was excluded from the final analysis due to suboptimal measurements. Therefore 14 participants in the cancer group and 15 participants in the control group were included in the analysis population.
Measure: Mean (95% Confidence Interval); unit: alpha units
Arm/Group | Cancer Group | Control Group
Number analyzed (Participants) | 14 | 15
alpha units
  Ampullary | .6968475 (.22) [.562102 to .831593] | .3483283 (.20) [.2318606 to .4647961]
  Distal 1 cm from ampullary | .7021826 (.35) [.4898464 to .9145189] | .4945491 (.28) [.3416003 to .647498]
  Distal periampullary | .4442996 (.15) [.3415441 to .5470551] | .4831275 (.17) [.3904288 to .5758262]
  Proximal 1 cm from ampulla | .6885187 (.29) [.5013549 to .8756826] | .4654624 (.34) [.2776132 to .6533117]
  Proximal periampullary | .4785118 (.22) [.3417855 to .6152382] | .43211449 (.33) [.2399311 to .6243588]
Statistical Analysis 1: Comparison: Cancer Group vs Control Group; Statistical significance p ≤ 0.05; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Mean Blood Vessel Radius (BVR)
Description: BVR serves as a marker for early increase of blood supply (EIBS).
Time Frame: Completion of study procedure (endoscopic ultrasound), approximately 30 minutes from procedure initiation
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Cancer Group | Control Group
Number analyzed (Participants) | 14 | 15
cm
  Ampullary | .003088 (.001) [.0022698 to .0039062] | .002035 (.001) [.0016118 to .0024582]
  Distal 1 cm from Ampulla | .0030272 (.001) [.0022997 to .0037547] | .0023467 (.001) [.0019386 to .0027548]
  Distal Periampullary | .002899 (.001) [.0021021 to .0036958] | .0024096 (.001) [.0021024 to .0027168]
  Proximal 1 cm from Ampulla | .0027802 (.001) [.0021426 to .0034178] | .0020825 (.001) [.0015238 to .0026411]
  Proximal Periampullary | .0023551 (.001) [.001627 to .0030832] | .0019793 (.001) [.0014618 to .0024968]
Statistical Analysis 1: Comparison: Cancer Group vs Control Group; Statistical significance p ≤ 0.05; Test type: Superiority or Other; p = 0.03, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Cancer Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 0/14 | 0/15

LIMITATIONS AND CAVEATS:
Small sample size, unmatched cohorts

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No